CLINICAL TRIAL: NCT04027426
Title: Families Becoming Healthy Together
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); The Miriam Hospital (Other); University of Memphis (Other); University at Buffalo (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Associate Dean of Research, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UTK IRB-18-04910-XP; 1R01DK121360 (NIH)
Record Dates: First submitted 2019-07-13; First posted 2019-07-22 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Childhood Obesity
Keywords: Habituation
MeSH Terms: conditions — Obesity; Pediatric Obesity; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blinded to randomization. Participants and providers will be blinded to study hypothesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FBT (family-based behavioral treatment) (Active Comparator): This condition will be prescribed the Traffic Light Diet (1000-1500 kcal/day, < 2 servings/day of RED [non-nutrient-dense, energy-dense] foods) and a > 60 min/day of MVPA prescription for children and > 30 min/day of MVPA for adults at least 5 days/week. FBT will receive a family-based, behavioral intervention to assist the targeted child and a participating adult caregiver with making changes in energy balance behaviors.
  Interventions: Behavioral: FBT
- FBT+Variety (Experimental): The FBT+Variety condition will receive FBT along with a limited variety prescription. In this prescription families will identify two RED foods, a dinner entree and snack food, and develop meal plans that reduce variety of RED foods by regularly consuming these foods and limiting consumption of other RED entrees and snack foods.
  Interventions: Behavioral: FBT+Variety

INTERVENTIONS:
Behavioral: FBT — FBT will receive a family-based, behavioral intervention for childhood obesity, consisting of group meetings once a week for months 1 to 4, twice a month for months 5 to 6, once a month for months 7 to 12, and once every two months for months 13 to 18 (29 sessions). For all meetings, the child and adult caregiver will be weighed and be provided with feedback, homework will be reviewed, and a behavioral lesson will be presented. At the 60-min meetings, the child and adult will attend separate 40 min group meetings, and then for the last 20 min of the meetings they will meet together with an individual therapist to address specific family-issues by developing behavioral action plans. No goals on variety in RED foods will be provided.
  Arms: FBT (family-based behavioral treatment)
Behavioral: FBT+Variety — This condition is FBT with a limited variety prescription. The limited variety prescription reduces the number of different RED foods consumed.
  Arms: FBT+Variety

SUMMARY:
The investigators plan to implement a novel limited RED (high-energy-dense) food variety prescription within a 18-month FBT to examine its effect on 18-month body mass index (BMI). This will be the first randomized control trial to examine how habituation rate, assessed via salivary habituation, mediates reduction in RED food intake, overall energy intake, and reductions in BMI over time, as well as if baseline habituation rate is a behavioral phenotype that moderates BMI outcomes. One hundred fifty-six children aged 8 to 12 years at > 85th percentile BMI will be randomized to one of two, 18-month interventions compared in our 6-month pilot study: FBT (family-based behavioral obesity treatment) or FBT+Variety. Child and adult caregiver assessments will occur at 0, 6, 12, and 18 months on anthropometrics, dietary intake (RED food variety, energy, and diet quality), habituation, and physical activity.

DETAILED DESCRIPTION:
Identifying successful methods for reducing long-term energy intake continues to be a challenge in obesity treatment. Basic behavioral research has found that the rate of habituation (i.e., rate of reduction in physiological and behavioral responding) to food is related to amount of food consumed, and faster habituation rates reduce food intake. The rate of habituation to food can be accelerated when variety in foods is limited, producing decreased intake. Thus, a dietary prescription that limits variety of high-energy-dense (HED) foods may boost ability to reduce long-term energy intake, enhancing long-term weight loss.

Furthermore, habituation rates to food show large individual variability. For example, individuals with overweight habituate slower to food than individuals with a healthy weight, and slower habituation rates predict greater increases in child standardized body mass index (ZBMI). Thus, slower habituation rates to food may be a behavioral phenotype for increased risk of suboptimal weight outcomes. Obesity interventions that accelerate habituation to food may then be more beneficial for those with this behavioral phenotype.

The investigators have been conducting a line of translational research that applies habituation theory to obesity treatment involving: 1) studies systematically testing basic concepts to better inform intervention development; 2) "proof-of-concept" testing; and 3) efficacy trials. The long-term goal of this research is to develop a dietary prescription that harnesses habituation as a mechanism for reducing long-term energy intake. This research has culminated in piloting a limited variety prescription (variety of both HED snack foods and entrees at dinner were limited) within a 6-month family-based behavioral obesity treatment (FBT) for children. Twenty-four families, with a child > 85th percentile BMI and aged 8 to 12 years, were randomized to FBT that included the Traffic Light Diet (1000-1500 kcal/day, < 2 servings/day of RED [HED] foods) and a > 60 min/day of moderate- to vigorous-intensity physical activity prescription or to FBT that included a limited dietary variety prescription (one RED snack food and dinner entrée were chosen; families regularly consumed these foods as compared to other RED snack foods and entrees) (FBT+Variety). At 6-months children in FBT+Variety had a significantly greater reduction in percent overweight than those in FBT (-15.4% vs.- 8.9%), and families in FBT+Variety had a lower daily intake of kcal from fat (351 kcal vs. 494 kcal). This limited dietary variety prescription shows promise for enhancing weight outcomes in FBT. However, research is needed to examine if limiting variety improves long-term weight loss, if this improvement is due to enhanced habituation, and explore if there is a behavioral phenotype that more greatly benefits from this dietary approach.

The investigators plan to implement a novel limited RED food variety prescription within an 18-month FBT to examine its effect on 18-month body mass index (BMI). This will be the first RCT to examine how habituation rate, assessed via salivary habituation, mediates reduction in RED food intake, overall energy intake, and reductions in BMI over time, as well as if baseline habituation rate is a behavioral phenotype that moderates BMI outcomes. One hundred fifty-six children aged 8 to 12 years at > 85th percentile BMI will be randomized to one of two, 18-month interventions compared in our 6-month pilot study: FBT or FBT+Variety. Child and adult caregiver assessments will occur at 0, 6, 12, and 18 months on anthropometrics, dietary intake (RED food variety, energy, and diet quality), habituation, and physical activity. The investigation was designed for all intervention sessions and assessments to be conducted in person. Due to COVID-19, modifications have occurred to the trial for health safety reasons. Initially, all meetings and assessments were to occur in-person. Due to the constant changing health safety requirements due to COVID-19, the trial puts in place health safety practices to maintain the safety of participants. Assessment meetings and program meetings will occur remotely via Zoom.

The primary aims are to determine for children:

1. Influence of FBT+Variety on long-term weight loss.
2. Influence of FBT+Variety on long-term habituation to RED foods. The habituation rate will mediate differences in dietary intake and BMI between conditions.

An exploratory aim is to examine in children:

1) Influence of habituation rate on moderating outcomes in FBT+Variety and FBT (identifying a behavioral phenotype that bests benefits from a limited variety prescription).

Comparisons will also be made between the conditions on all child dietary and activity measures. Additionally, adult caregiver measures will be examined, with outcomes anticipated to be similar to child outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age between 8 and 12 years
* > 85th percentile BMI
* one adult caregiver (> 18 years) living in the household with a BMI > 25 kg/m2 willing to attend treatment meetings

Exclusion Criteria:

* child and adult caregiver report living in two separate households for > 2 days per week
* child or adult caregiver report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q) (individuals reporting joint problems, prescription medication usage, or other medical conditions that could limit exercise will be required to obtain written physician consent to participate)
* child or adult caregiver report being unable to walk for 2 blocks (1/4 mile) without stopping
* child or adult caregiver report major psychiatric diseases or organic brain syndromes
* child or adult caregiver report currently participating in a weight loss program and/or taking weight loss or appetite regulation medication or lost > 5% of body weight during the past 6 months
* child report having bariatric surgery for weight loss/planning to have bariatric surgery in the next 18 months, adult caregiver having bariatric surgery in the previous two years or planning to have bariatric surgery in the next 18 months
* adult caregiver reports being pregnant, lactating, less than 6 months post-partum or plans to become pregnant in the next 18 months
* child or adult caregiver report planning to move outside of the metropolitan area (defined as from Nashville to the east state border of Tennessee) or Memphis (this may include residents who live in Arkansas or Mississippt) within the time frame of the investigation
* child or adult caregiver report dietary restrictions for medical reasons
* child or adult caregiver report allergies to lemon or lime juice (used in habituation measures)
* child is not able to read at a third-grade reading level.
* do not have reliable internet access.
* participation in the study creates conflict with child's educational support or health condition treatment/program due to time needs, incompatible goals, or strain on family resources.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Child and adult body mass index | Change from 0 to 6, and 6 to 18 months
  Child's and adult caregiver's weight will be assessed by an electronic scale and height will be measured by a stadiometer.
Child and adult salivary habituation | Change from 0 to 6, and 6 to 18 months
  To assess habituation of salivary responses to food cues, whole mouth parotid salivary flow will be measured using the Strongin-Hinsie Peck method. Two measures will be taken, one with juice and one with food.

SECONDARY OUTCOMES:
Child and adult dietary Intake | Change from 0 to 6, and 6 to 18 months
  Dietary intake for both the child and adult caregiver will be assessed by 3 (2 weekdays and 1 weekend day) 24-hour dietary phone recalls, using the five-step, multiple-pass method. Variables of interest will be the variety of RED foods consumed over the three days; and the mean over the three days of daily servings and kcal from RED foods, kcal, energy density (kcal/g), and Healthy Eating Index (HEI)-2015. Adherence to the prescriptions in the two conditions will be examined. At 6, 12, and 18 months, the percentage of goals met each day will be calculated, with a mean percentage calculated. We will also provide a detailed list of snack foods to participants, and they will be asked to indicate which of the foods on the list were eaten during the previous month, regardless of quantity consumed.
Child and adult physical activity via wGT3X-BT | Change from 0 to 6, and 6 to 18 months
  The wGT9x (ActiGraph, LLC, Pensacola, FL) will objectively measure time spent in MVPA (physical activity at > 3.0 metabolic equivalents units).
Child percent overweight | Change from 0 to 6, and 6 to 18 months
  Percent overweight (%OW) will also be calculated (100*[BMI/50th percentile BMI for child age and sex]).
Child and adult waist circumference | Change from 0 to 6, and 6 to 18 months
  Waist circumference (WC) will be measured using standard procedures.
Meal planning, preparation, and grocery shopping | Change from 0 to 6, and 6 to 18 months
  Parent time scarcity and fatigue as barriers to planning and preparing meals will measure frequency of occurrence of these barriers.
Child eating pathology | Change from 0 to 6, and 6 to 18 months
  Child eating pathology will be assessed using the Kid's Eating Disorder Survey
Home Food Inventory | Change from 0 to 6, and 6 to 18 months
  Self-reported inventory of foods available in the household will be assessed
Child and Adult Sleep Habits | Change from 0 to 6, and 6 to 18 months
  Usual sleeping and waking time will be collected
Child Routines | Change from 0 to 6, and 6 to 18 months
  Parent-report measure of commonly occurring routines in school-aged children will measure the frequency of occurrence of routines in children.
Compliance and process data | 6, 12, and 18 months
  Total number of weekly, and type, of self-monitoring records (hard copy or electronic) completed will be assessed. Number of treatment sessions attended will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Hollie Raynor, PhD RD LDN, Principal Investigator — University of Tennessee Knoxville
Locations (1):
- Healthy Eating and Activity Lab, University of Tennessee, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altman M, Wilfley DE. Evidence update on the treatment of overweight and obesity in children and adolescents. J Clin Child Adolesc Psychol. 2015;44(4):521-37. doi: 10.1080/15374416.2014.963854. Epub 2014 Dec 12. PMID 25496471
- [Background] Epstein LH, Temple JL, Roemmich JN, Bouton ME. Habituation as a determinant of human food intake. Psychol Rev. 2009 Apr;116(2):384-407. doi: 10.1037/a0015074. PMID 19348547
- [Background] Epstein LH, Robinson JL, Temple JL, Roemmich JN, Marusewski AL, Nadbrzuch RL. Variety influences habituation of motivated behavior for food and energy intake in children. Am J Clin Nutr. 2009 Mar;89(3):746-54. doi: 10.3945/ajcn.2008.26911. Epub 2009 Jan 28. PMID 19176724
- [Background] Temple JL, Giacomelli AM, Roemmich JN, Epstein LH. Dietary variety impairs habituation in children. Health Psychol. 2008 Jan;27(1S):S10-9. doi: 10.1037/0278-6133.27.1.S10. PMID 18248101
- [Background] Epstein LH, Fletcher KD, O'Neill J, Roemmich JN, Raynor H, Bouton ME. Food characteristics, long-term habituation and energy intake. Laboratory and field studies. Appetite. 2013 Jan;60(1):40-50. doi: 10.1016/j.appet.2012.08.030. Epub 2012 Oct 22. PMID 23085682
- [Background] Epstein LH, Robinson JL, Temple JL, Roemmich JN, Marusewski A, Nadbrzuch R. Sensitization and habituation of motivated behavior in overweight and non-overweight children. Learn Motiv. 2008 Aug;39(3):243-255. doi: 10.1016/j.lmot.2008.03.001. PMID 19649135
- [Background] Bond DS, Raynor HA, McCaffery JM, Wing RR. Salivary habituation to food stimuli in successful weight loss maintainers, obese and normal-weight adults. Int J Obes (Lond). 2010 Mar;34(3):593-6. doi: 10.1038/ijo.2009.267. Epub 2009 Dec 15. PMID 20010900
- [Background] Bond DS, Raynor HA, Vithiananthan S, Sax HC, Pohl D, Roye GD, Ryder BA, Wing RR. Differences in salivary habituation to a taste stimulus in bariatric surgery candidates and normal-weight controls. Obes Surg. 2009 Jul;19(7):873-8. doi: 10.1007/s11695-009-9861-3. Epub 2009 May 20. PMID 19455371
- [Background] Epstein LH, Carr KA, Cavanaugh MD, Paluch RA, Bouton ME. Long-term habituation to food in obese and nonobese women. Am J Clin Nutr. 2011 Aug;94(2):371-6. doi: 10.3945/ajcn.110.009035. Epub 2011 May 18. PMID 21593492
- [Background] Temple JL, Giacomelli AM, Roemmich JN, Epstein LH. Overweight children habituate slower than non-overweight children to food. Physiol Behav. 2007 Jun 8;91(2-3):250-4. doi: 10.1016/j.physbeh.2007.03.009. Epub 2007 Mar 16. PMID 17459429
- [Background] Aspen VA, Stein RI, Wilfley DE. An exploration of salivation patterns in normal weight and obese children. Appetite. 2012 Apr;58(2):539-42. doi: 10.1016/j.appet.2011.11.027. Epub 2011 Dec 3. PMID 22172456
- [Background] Epstein LH, Kilanowski C, Paluch RA, Raynor H, Daniel TO. Reducing variety enhances effectiveness of family-based treatment for pediatric obesity. Eat Behav. 2015 Apr;17:140-3. doi: 10.1016/j.eatbeh.2015.02.001. Epub 2015 Feb 13. PMID 25706950

DOCUMENTS (1):
  • Informed Consent Form (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT04027426/ICF_009.pdf